CLINICAL TRIAL: NCT02367534
Title: Islet Transplantation Through an Indwelling Catheter in the Umbilical Vein
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Principal Investigator, Jianming Tan, Director, Organ transplantation intitute, Fuzhou General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Umbilical-vein
Record Dates: First submitted 2015-01-23; First posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Umbilical vein (Experimental): umbilical vein catheterization
  Interventions: Procedure: umbilical vein catheterization

INTERVENTIONS:
Procedure: umbilical vein catheterization — A 7 cm incision was made in the middle-right of upper abdominal. The umbilical vein was identified located 4cm beyond umbilicus, which was then half dissected transversely and the atresic venous lumen was recanalized with a common duct probe (3mm-5mm, BAKES). A breakthrough feeling would be sensed after approaching forward for 10-14cm and the umbilical vein was successfully recanalized. The common duct probe was pulled out. A catheter (single lumen central venous catheter, 16-20G, TUOREN, China) was then cannulated for 15cm into left branch of portal vein through umbilical vein. The procedure was observed with Doppler ultrasound (LOGIQ S6, GE).

SUMMARY:
Islet transplantation is one of the effective and promising options for type 1 diabetes mellitus treatment1-4. The liver is the primary target location for infusion and portal vein catheterization is generally used. Percutaneous transjugular, percutaneous transhepatic, laparoscopically transmesenteric and laparoscopically transumbilical approaches were often utilized to access the portal. Current islet infusion approach via portal vein of liver has various defects. Percutaneous trans-hepatic puncture is risk of possible severe hemorrhage and portal thrombosis. The laparoscopic entry techniques require longer surgical duration and have an increased rate of catheterization failure. Moreover, the catheters were not allowed to indwell for subsequent infusions.

In the current study, the investigators aim to performed open surgery, catheterized the umbilical vein and infused islets into the portal vein. The catheter was indwelled for one month after surgery. Therapeutic effects, surgical parameters and complications were observed to evaluate feasibility and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 to 60 years of age.
* Ability to provide written informed consent.
* Clinical history compatible with type 1 diabetes (T1DM) as defined by the WHO guidelines(2007) on the Diagnosis and classification of Diabetes Mellitus.
* manifest signs and symptoms that are severe enough to be incapacitating.
* Basal C-peptide<0.5ng/mL
* patients with poor diabetes control (HbA1c >7% but <12%)
* progressive diabetic complications.

Exclusion Criteria:

* age <18 years or >60 years
* diabetic history <5 years
* BMI>27
* body weight >80kg
* exogenous insulin requirement >1 unit/kg/day
* severe anemia (male <8g/dl, female <7g/dl)
* low white blood cell count (<3000/dl)
* liver dysfunction
* Symptomatic peptic ulcer disease
* Any malignancy
* Active infection including hepatitis B, hepatitis C, HIV, or TB
* panel reactive antibody >20%
* Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
hemorrhage | 1 month

SECONDARY OUTCOMES:
Infection | 6 month
Exogenous insulin requirement | 1 year
Glucose | 1 year
C-peptide | 1 year